CLINICAL TRIAL: NCT03790267
Title: Functional Outcomes and Quality of Life Reported by Adult Patients Undergoing Elective Hip, Knee and Shoulder Arthroplasty
Brief Title: Functional Outcomes and Quality of Life in Hip, Knee and Shoulder Arthroplasty
Acronym: PaRIS-IOR
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor of Orthopaedics, Istituto Ortopedico Rizzoli
Other Study IDs: PaRIS-IOR
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hip arthroplasty
  Interventions: Other: Questionnaire administration
- Knee arthroplasty
  Interventions: Other: Questionnaire administration
- Shoulder arthroplasty
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — One questionnaire (Euro Quality 5 Dimensions, EQ-5D) for the general assessment of patient's health status will be administered to all the patients in the study. One joint-specific questionnaires will be administered to patients depending on the surgery procedure they will be undergoing. Hip disability and Osteoarthritis Outcome Score - Short Form (HOOS-PS) for patients undergoing hip replacement (6); Knee injury and Osteoarthritis Outcome Score - Short Form (KOOS-PS) for patients undergoing knee replacement (7); the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES), for patients undergoing shoulder implants.

SUMMARY:
PaRIS-IOR is a prospective observational study that aims to collect and analyze functional outcomes and quality of life reported by patients undergoing elective hip, knee and shoulder arthroplasty at the IRCCS Rizzoli Orthopedic Institute (IOR).

DETAILED DESCRIPTION:
PaRIS-IOR is a prospective observational study that aims to collect and analyze functional outcomes and quality of life reported by patients undergoing elective hip, knee and shoulder arthroplasty at the IRCCS Rizzoli Orthopedic Institute (IOR). IOR was selected as a pilot center for the launch of the OECD's PaRIS Initiative in Italy, whose purpose is to accelerate the adoption and reporting of validated, standardised, internationally-comparable patient-reported indicators, particularly within patient registries.

PaRIS-IOR's study population will consist of consecutive patients undergoing hip, knee and shoulder arthroplasty performed at 6 Operative Units of the IOR. The study will last 30 months and will include a 12-month recruitment period, a 12-month follow-up and 6 months for data analysis and reporting. Functional outcomes and quality of life will be detected through the administration of validated questionnaires (EQ-5D, HOOS, KOOS, ASES). The questionnaires will be administered in the month preceding the surgical procedure in the clinic or in the ward, while the 2 follow-up questionnaires will be send by mail at patients' home. The collected data will be combined with those routinely collected by the Registry of Orthopedic Prosthetic Implantology (RIPO), already active at the IOR since year 1990.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-95 years
2. Be on the list for an elective primary arthroplasty of hip, knee or shoulder
3. Availability to sign the informed consent

Exclusion Criteria:

1. Severe cognitive impairment
2. To be listed for arthroplasty for musculoskeletal cancer
3. Not eligible for the surgical intervention

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutive patients undergoing hip, knee and shoulder arthroplasty. Patients will be enrolled at 6 operative units of the IOR (Orthopedic and Traumatological I Clinic, Orthopedic and Traumatological Clinic II, Orthopedic and Traumatologic Clinic III, Reconstructive Orthopedic Surgery - Innovative Techniques / Revision surgery of hip prosthesis and new implant development, Surgery of the Shoulder and Elbow, Orthopedics-Traumatology and Prosthetic Surgery and of hip and knee replanting). For patients accessing through the "hospitalization-before-surgery" pathway, the enrollment will take place in the specific ambulatory in the month preceding the intervention. The remaining patients will be enrolled directly at the operative Units involved.
Sampling Method: Non-Probability Sample
Enrollment: 4260 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Functional outcomes: total score of the joint-specific functional scales. | Baseline
  The joint-specific functional scales derive from the following validated questionnaires: Hip disability and Osteoarthritis Outcome Score - Short Form (HOOS-PS) for patients undergoing hip replacement; Knee injury and Osteoarthritis Outcome Score - Short Form (KOOS-PS) for patients undergoing knee replacement; the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES), for patients undergoing shoulder implants. For all questionnaires the items are coded from 0 to 4, no functional difficulty to extreme functional difficulty respectively. The total score of the questionnaires can go from 0 (worst outcome) to 100 (best outcome).
Functional outcomes: total score of the joint-specific functional scales. | 6 months after surgery
  The joint-specific functional scales derive from the following validated questionnaires: Hip disability and Osteoarthritis Outcome Score - Short Form (HOOS-PS) for patients undergoing hip replacement; Knee injury and Osteoarthritis Outcome Score - Short Form (KOOS-PS) for patients undergoing knee replacement; the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES), for patients undergoing shoulder implants. For all questionnaires the items are coded from 0 to 4, no functional difficulty to extreme functional difficulty respectively. The total score of the questionnaires can go from 0 (worst outcome) to 100 (best outcome).
Functional outcomes: total score of the joint-specific functional scales. | 12 months after surgery
  The joint-specific functional scales derive from the following validated questionnaires: Hip disability and Osteoarthritis Outcome Score - Short Form (HOOS-PS) for patients undergoing hip replacement; Knee injury and Osteoarthritis Outcome Score - Short Form (KOOS-PS) for patients undergoing knee replacement; the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES), for patients undergoing shoulder implants. For all questionnaires the items are coded from 0 to 4, no functional difficulty to extreme functional difficulty respectively. The total score of the questionnaires can go from 0 (worst outcome) to 100 (best outcome).
Euro-Quality-5-Dimensions questionnaire scores. | Baseline
  Euro Quality 5 Dimensions, EQ-5D, will be used for the general assessment of patient's health status. The EQ-5D is a standardized instrument for measuring generic health status. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents are asked to choose one of the statements which best describes their health status of surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Euro-Quality-5-Dimensions questionnaire scores. | 6 months after surgery
  Euro Quality 5 Dimensions, EQ-5D, will be used for the general assessment of patient's health status. The EQ-5D is a standardized instrument for measuring generic health status. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents are asked to choose one of the statements which best describes their health status of surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Euro-Quality-5-Dimensions questionnaire scores. | 12 months after surgery
  Euro Quality 5 Dimensions, EQ-5D, will be used for the general assessment of patient's health status. The EQ-5D is a standardized instrument for measuring generic health status. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents are asked to choose one of the statements which best describes their health status of surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Visual analogue scale (EQ-VAS) scores | Baseline
  The respondents evaluate their overall health status using the visual analogue scale (EQ-VAS), asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100: (0) corresponds to " the worst health you can imagine", and (100) corresponds to "the best health you can imagine".
Visual analogue scale (EQ-VAS) scores | 6 months after surgery
  The respondents evaluate their overall health status using the visual analogue scale (EQ-VAS), asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100: (0) corresponds to " the worst health you can imagine", and (100) corresponds to "the best health you can imagine".
Visual analogue scale (EQ-VAS) scores | 12 months after surgery
  The respondents evaluate their overall health status using the visual analogue scale (EQ-VAS), asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100: (0) corresponds to " the worst health you can imagine", and (100) corresponds to "the best health you can imagine".

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Derived] Golinelli D, Grassi A, Tedesco D, Sanmarchi F, Rosa S, Rucci P, Amabile M, Cosentino M, Bordini B, Fantini MP, Zaffagnini S. Patient reported outcomes measures (PROMs) trajectories after elective hip arthroplasty: a latent class and growth mixture analysis. J Patient Rep Outcomes. 2022 Sep 9;6(1):95. doi: 10.1186/s41687-022-00503-5. PMID 36085337
- [Derived] Grassi A, Golinelli D, Tedesco D, Rolli M, Bordini B, Amabile M, Rucci P, Fantini MP, Zaffagnini S. Patient-reported outcome measures (PROMs) after elective hip, knee and shoulder arthroplasty: protocol for a prospective cohort study. BMC Musculoskelet Disord. 2019 Aug 15;20(1):374. doi: 10.1186/s12891-019-2745-3. PMID 31416443

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT03790267/Prot_SAP_001.pdf